CLINICAL TRIAL: NCT07000591
Title: The Effect of Massage Based on the Human Caring Model on Self-Efficacy, Symptom Management, and Caregiver Burden in Patients With Epilepsy: A Randomized Controlled Trial
Brief Title: Massage Based on the Human Caring Model in Epilepsy
Acronym: Massage Based
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Muş Alparslan University (Other)
Collaborators: Scientific Research Projects (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MAUN-SBF-CO-01
Record Dates: First submitted 2025-05-24; First posted 2025-06-03 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-05

CONDITIONS: Epilepsy
Keywords: Epilepsy; Human Caring Model; Self-Efficacy; Symptom Management
MeSH Terms: conditions — Epilepsy | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: In this clinical trial, Jean Watson's Human Caring Model will be used. The model provides a holistic and humane approach to care, addressing patients' physical, emotional, and spiritual needs. Interventions based on Watson's "Caring" approach aim to promote patient relaxation, build a sense of security, and improve quality of life. Thus, the healing effect of nursing care during the treatment process will be supported.
Masking Description: Due to the nature of the study, blinding was not performed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): After the initial data is collected, no interventions other than routine nursing care will be applied to the patients and their caregivers. Not intervening in the control group will be necessary to accurately evaluate whether the research hypothesis is significant. This approach will ensure that only the effects of the intervention are isolated, allowing for a proper analysis of the differences between groups based on the research hypothesis. For this group, the researchers will administer the "Patient Introduction Form," the "Epilepsy Self-Efficacy Scale," and the "Epilepsy Symptom Management Scale" to the patients, and the "Caregiver Introduction Form" and the "Zarit Burden Interview" to the caregivers, as data collection tools, eight weeks after the initial assessment to collect the final test data.
- Experimental group (Experimental): Patients will receive a neck massage based on Watson's Human Caring Model in addition to standard medical care. The massage will be performed three times a week for eight weeks, totaling 24 sessions. Sessions will last 30 minutes and follow evidence-based nursing interventions. Care will be individualized and delivered in a calming environment.
  Pre- and post-intervention assessments will include the Epilepsy Self-Efficacy Scale and the Epilepsy Symptom Management Scale for patients, and the Zarit Burden Interview for caregivers. Caregivers will also complete an introductory form. All data will be collected at baseline and after eight weeks. The massage's impact on both patient outcomes and caregiver burden will be evaluated.
  Interventions: Other: Experimental Group

INTERVENTIONS:
Other: Experimental Group — Patients will receive a neck massage based on Watson's Human Caring Model in addition to standard medical care. The massage will be performed three times a week for eight weeks, totaling 24 sessions. Sessions will last 30 minutes and follow evidence-based nursing interventions. Care will be individualized and delivered in a calming environment.
  Pre- and post-intervention assessments will include the Epilepsy Self-Efficacy Scale and the Epilepsy Symptom Management Scale for patients, and the Zarit Burden Interview for caregivers. Caregivers will also complete an introductory form. All data will be collected at baseline and after eight weeks. The massage's impact on both patient outcomes and caregiver burden will be evaluated.
  Other Names: Treatment
  Arms: Experimental group

SUMMARY:
This randomized controlled study will be conducted with 96 epilepsy patients and their caregivers at Atatürk University Research Hospital between November 2024 and February 2026. Participants will be randomly assigned to experimental and control groups. The experimental group will receive neck massage based on Jean Watson's Human Caring Model three times a week for eight weeks. Data will be collected using various scales to evaluate self-efficacy, symptom management, and caregiver burden before and after the intervention.

DETAILED DESCRIPTION:
This study will be conducted between November 15, 2024, and February 15, 2026, at Atatürk University Research Hospital in Erzurum. The population will consist of patients diagnosed with Generalized Tonic-Clonic Seizures or Focal Epilepsy. The sample size will be determined using a priori power analysis, and a total of 96 participants, including 48 patients in each group, will be included in the study along with their caregivers. Participants will be randomly assigned to the experimental and control groups using a simple randomization method via random.org. Data collection tools will include the Patient and Caregiver Information Forms, Epilepsy Self-Efficacy Scale, Zarit Caregiver Burden Scale, Epilepsy Symptom Management Scale, and Neck Massage Follow-Up Form. Patients in the experimental group will receive neck massage based on the Human Caring Model three times a week for eight weeks, for a total of 24 sessions. Participants will be informed before each massage session, and the procedures will be conducted according to a standardized protocol. Pre- and post-massage assessments will be conducted to monitor changes in symptom management, self-efficacy levels, and caregiver burden. Jean Watson's Human Caring Model will be used as the theoretical framework throughout the entire process.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years,
* Diagnosed with Generalized Tonic-Clonic Seizures or Focal Epilepsy,
* Able to speak and understand Turkish,
* Conscious and alert,
* Able to communicate verbally,
* No history of neck trauma,
* No cervical disc herniation,
* No severe headaches or migraines,
* Not diagnosed with cancer,
* No neurological and/or psychiatric disorders affecting cognitive function,
* No acute (recently developed) health issues (e.g., heart attack, fainting),
* No uncontrolled high blood pressure,
* No use of analgesic medications in the past 24 hours,
* No contraindications to massage therapy (e.g., advanced COPD, asthma, heart or kidney failure, malignant conditions, febrile illnesses, or pregnancy),
* No skin issues (rash, redness, lesions, heat increase, swelling, edema, bone abnormalities, or localized infections) in the area where massage is to be applied.

Exclusion Criteria

* Declining to continue participation in the study,
* Experiencing pain during massage application,
* Changes in the pharmacological treatment regimen,
* Failing to attend massage sessions,
* Development of undesirable effects (e.g., bruising or discoloration) in the massage area, which leads to termination of sessions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2025-06-15 (Actual); Primary Completion 2025-06-15 (Actual); Study Completion 2025-09-15 (Actual)

PRIMARY OUTCOMES:
Epilepsy Self-Efficacy Scale | four months
  The Epilepsy Self-Efficacy Scale was originally developed by DiIorio et al. in 1992 as a 25-item tool to assess individuals' belief in their ability to manage their epilepsy. In 2000, 8 additional items were included in the original scale. The Turkish validity and reliability study was conducted in 2019 by Öznur Adadıoğlu. Cronbach's alpha values were reported as 0.88 for the management factor, 0.84 for the general management factor, 0.82 for illness and medication management, 0.55 for seizure management, and 0.91 for the total scale. Based on factor analysis, 2 items were removed, and the final Turkish version included 31 items. Items are scored from "0 - I cannot do at all" to "10 - I am absolutely sure I can do," and total scores range from 0 to 310. When averaged, scores range from 0 to 10. Higher scores indicate greater self-efficacy.
Zarit Burden Interview (ZBI) | four months
  The Zarit Burden Interview was developed in 1980 by Zarit, Reever, and Bach-Peterson to assess the level of stress experienced by caregivers. It consists of 22 items addressing social and emotional aspects of caregiving. Each item is scored on a 5-point Likert scale ranging from "never" to "nearly always." Total scores range from 0 to 88, with higher scores indicating greater caregiver burden. Reliability studies found internal consistency coefficients between 0.87 and 0.94. The Turkish validity and reliability study was conducted by İnci in 2006, with a Cronbach's alpha of 0.95.
Epilepsy Symptom Management Scale | four months
  This scale was developed by the researchers based on relevant literature (Kurt & Ünsar, 2009; Yeşilbalkan et al., 2008; Yıldırım et al., 2011; Tülek et al., 2016; Mollaoğlu et al., 2015; Önsöz & Usta Yeşilbalkan, 2013; Atay Turan et al., 2007) for use in a doctoral dissertation. Initially, 40 items were drafted. Following expert review, two items were removed, one was split into two, and six were revised, resulting in a final version with 39 items. The scale provides a holistic, user-friendly tool for epilepsy patients to self-assess all symptoms in a single form. Patients indicate whether they experienced symptoms in the past week (Yes/No). If "Yes," they rate the impact on a 5-point Likert scale: 1 = Not at all disturbing to 5 = Extremely disturbing. Total scores range from 0 to 195, with higher scores indicating greater symptom burden. To assess content validity, 10 experts evaluated each item using Davis' method, which involves rating items as: 1 = Not appropriate, 2 = Needs major

CONTACTS AND LOCATIONS:
Locations (1):
- Atatürk University, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No